CLINICAL TRIAL: NCT05951023
Title: Endotype-Targeted Therapy to Rescue OSA Patients Struggling With CPAP Adherence (TOP-CPAP): a Pilot Trial
Brief Title: Endotype-Targeted Therapy to Rescue OSA Patients Struggling With CPAP Adherence (TOP-CPAP)
Acronym: TOP-CPAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: American Academy of Sleep Medicine (Other)
Responsible Party: Principal Investigator, Christopher Schmickl, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 190560; 277-JF-22 (Other Grant/Funding Number: American Academy of Sleep Medicine Foundation (AASMF))
Record Dates: First submitted 2023-06-17; First posted 2023-07-18 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; OSA; Continuous Positive Airway Pressure; CPAP; Adherence; Eszopiclone; Endotype; Arousal Threshold
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Eszopiclone

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eszopiclone (Experimental): Subjects will be asked to take their study drugs nightly at bedtime and use their CPAP during sleep as much as possible
  Interventions: Drug: Eszopiclone 2 mg
- Placebo (Placebo Comparator): Subjects will be asked to take their study drugs nightly at bedtime and use their CPAP during sleep as much as possible
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eszopiclone 2 mg — Eszopiclone tablet (encapsulated)
  Other Names: Lunesta
  Arms: Eszopiclone
Drug: Placebo — Sugar capsule manufactured to match encapsulated Eszopiclone
  Arms: Placebo

SUMMARY:
More than 10% of the US population have obstructive sleep apnea (OSA). Standard of care is therapy with CPAP (continuous positive airway pressure) which virtually eliminates OSA. However, most patients use CPAP only for part of the night (4-5hours) and about 50% patients discontinue CPAP long-term. Alternative therapies are limited, thus many OSA patients remain at risk of OSA sequelae (e.g. sleepiness, memory issues, high blood pressure, etc.). Importantly, different patients get OSA for different reasons, and recent data show that some of the underlying causes of OSA ("endotypes") such as having a low arousal threshold (i.e. waking up easily) are associated with lower CPAP adherence. Using a randomized controlled trial design, this will be the first study using a targeted intervention to manipulate the underlying OSA causes (i.e., giving a safe hypnotic to patients with OSA to increase the arousal threshold) to test the hypothesis that endotype-targeted therapy increases CPAP-adherence in patients who have low but continued CPAP usage. Ultimately, this strategy may improve the care and outcomes of millions of undertreated OSA patients.

DETAILED DESCRIPTION:
This double-blind, randomized, placebo-controlled, single-center, phase II trial, will test if endotype-targeted drug therapy increases CPAP adherence. Patients with low CPAP adherence (i.e. CPAP use 0.5-4h/night) will be randomized in parallel to CPAP+Eszopiclone vs CPAP+Placebo for 2 weeks. The primary outcome is mean TimeOnCPAP/night on days 2-14 after initiation of study drugs.

Aim 1: To test the effect of eszopiclone on CPAP usage in unselected OSA patients with low CPAP adherence.

Hypothesis 1: Eszopiclone improves CPAP usage more than placebo.

Aim 2: To test the effect of eszopiclone on CPAP usage in OSA patients with a low vs a high arousal threshold (ArTH) endotype.

Hypothesis 2: Eszopiclone improves CPAP usage substantially more in OSA patients with a low vs a high ArTH.

Further, this study will explore the mechanisms through which eszopiclone may affect CPAP usage, the effect of eszopiclone on underlying sleep apnea severity, and if the intervention and its potential effects on adherence translate into changes in clinically important outcomes (i.e., vigilance and sleepiness).

ELIGIBILITY:
Inclusion Criteria:

* Ages 21-65 years old
* Body Mass Index <32 kg/m^2
* Physician diagnosis of OSA (AHI ≥ 10) based on a clinical sleep study within the past 2 years (subjects who report a history of sleep apnea but do not have a sleep study report from the past 2 years available will be offered an overnight home sleep apnea test to verify OSA diagnosis)
* AHI>5/h on the overnight research sleep study #1
* Subject had the opportunity to use CPAP for at least 1 month
* Continuous positive airway pressure (CPAP) data can be queried remotely and shows usage 0.5-4h/night (based on most recent 30 day period)
* Interest to continue trying CPAP

Exclusion Criteria:

* "SAVE CPAP Side Effect Score" >3 (1 point for each: dry mouth, nasal symptoms, CPAP pressure intolerance, claustrophobia, noise problems, soreness/skin irritation, mask fit/leak problems)
* Any high-risk features: Epworth sleepiness score ≥18, safety-critical profession (e.g., commercial driver), prior sleep-related car accident, substantial hypoxemia during sleep [SpO2<70% for >5min] or awake [SpO2<92%]
* Any uncontrolled medical/psychiatric condition, or safety concern based on MD judgment
* Pregnancy/Breastfeeding (current or planned during the next month)
* Inability to complete study procedures, such as questionnaires that are only available/validated in English
* Other known untreated sleep fragmenting disorder, such as periodic limb movement disorder, or narcolepsy
* Unwilling or unable to withhold CPAP during polysomnography
* Presence of tracheostomy
* Hospitalization within the past 90 days
* Allergy to the study drug
* Regular use of opioids, or benzodiazepines
* Chronically using study drug or other hypnotic
* Significant circadian rhythm disorder or sleepwalking as an adult
* Active illicit substance use or >3 oz nightly alcohol use
* Prisoners
* Cognitive impairment, unable to provide consent, or unable to carry out research procedures
* Safety concern based on MD judgment

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Mean use per night of continuous positive airway pressure (CPAP) | days 2-14 after initiation of study drugs
  Based on device recorded usage

SECONDARY OUTCOMES:
Alternative measures of CPAP usage | days 2-14 after initiation of study drugs
  E.g. percentage of nights with CPAP >4h
Response Speed | days 2-14 after initiation of study drugs
  Based on 10-minute Psychomotor vigilance task (PVT)
Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance (SDA) instrument | days 2-14 after initiation of study drugs
  Based on response pattern scoring, the PROMIS 8-item SDA score will be converted into a T-score with a mean of 50 (reflecting the average for the United States general population) and a standard deviation of 10. Higher t-scores reflect greater sleep disturbance.
Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep-Related Impairment (SRI) instrument | days 2-14 after initiation of study drugs
  Based on response pattern scoring, the PROMIS 8-item SRI score will be converted into a T-score with a mean of 50 (reflecting the average for the United States general population) and a standard deviation of 10. Higher t-scores reflect greater sleep-related impairment.
Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue instrument | days 2-14 after initiation of study drugs
  Based on response pattern scoring, the PROMIS 8-item Fatigue score will be converted into a T-score with a mean of 50 (reflecting the average for the United States general population) and a standard deviation of 10. Higher t-scores reflect greater sleep-related impairment.
Epworth Sleepiness Scale (ESS) | days 2-14 after initiation of study drugs
  The ESS is an 8-item instrument assessing the likelihood of dozing off in 8 different situations with points for each item ranging from 0 to 3 (0 = would never doze off; 3 = high chance of dozing off). The points for each item are summed up, thus the total score ranges from 0 to 24, with higher ESS scores indicating greater sleepiness.
Apnea Hypopnea Index | day1 of study drugs
  The AHI is a measure of sleep apnea severity and is defined as the number of apneas and hypopneas per hour of sleep.
Mean Blood Pressure (mmHg) | day 14 after initiation of study drugs
  Average of two in-office blood pressure measurements

OTHER OUTCOMES:
Sleep Apnea Traits with special focus on arousal threshold | day1 of study drugs
  Quantified from routine polysomnography data.
Average total sleep time per night | days 2-14 after initiation of study drugs
  Based on actigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Christopher N Schmickl, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- UC San Diego; Altman Clinical and Translational Research Institute Building, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No